CLINICAL TRIAL: NCT02627014
Title: Effect of Treatment of Temporomandibular Joint in Patients With Chronic Migraine and Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Eva Segura Ortí (PhD), Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CM_TMD_1
Record Dates: First submitted 2015-12-04; First posted 2015-12-10 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Chronic Migraine; Temporomandibular Disorders
Keywords: Chronic Migraine; Temporomandibular Disorders; Physical Therapy; Manual Therapy; Home physical Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INTERVENTION (Experimental): Manual Therapy in temporomandibular joint and cervical region. Home physical therapy in temporomandibular joint and cervical region.
  Interventions: Other: Manual therapy; Other: Home physical therapy
- CONTROL (Active Comparator): Manual therapy in cervical region Home physical therapy in cervical region
  Interventions: Other: Manual therapy in cervical region; Other: Home physical therapy in cervical region

INTERVENTIONS:
Other: Manual therapy — 6 treatments: 2 treatments for week
  1 treatment = 30 minutes
  Arms: INTERVENTION
Other: Home physical therapy — once a day: 15 minutes
  Arms: INTERVENTION
Other: Manual therapy in cervical region — 6 treatments: 2 treatments for week
  1 treatment = 30 minutes
  Arms: CONTROL
Other: Home physical therapy in cervical region — once a day: 15 minutes
  Arms: CONTROL

SUMMARY:
The aim of this study is to determine whether treatment of temporomandibular joint is more effective than usual care in patients with chronic migraine and temporomandibular disorders to reduce pain.

DETAILED DESCRIPTION:
The aim of this study is to determine whether treatment of temporomandibular joint added to the control group treatment and drug therapy patient base is more effective than just using the control group treatment and drug therapy in patients with chronic migraine and temporomandibular disorders to reduce pain and improve the quality of life related to health of patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine (ICHD_III beta, 2013)
* Temporomandibular disorders (RDC/TMD)

Exclusion Criteria:

* other neurological disease
* psychiatric diseases
* Physical therapy treatment in the last 6 months
* dental treatment in the last 6 months
* surgery or trauma in the orofacial region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Headache Impact Test (HIT-6) | 3 months

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 3 months
Quality of life (SF-36) | 3 months
Sleep Quality | 3 months
  Pittsburgh Sleep Quality Index
Pain threshold pressure | 3 months
  Pressure algometer in masticatory muscle (area trigeminal) and control point in area extra-trigeminal
Pain catastrophizing scale (PCS) | 3 months
Craniofacial Pain and Disability Inventory (CF-PDI) | 3 months
Tampa scale of Kinesiophobia (TSK) | 3 months
Tampa scale of Kinesiophobia of cranio-mandibular disorder (TSK-TCM) | 3 months
Maximal Mouth Opening pain free | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Garrigós, Principal Investigator — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Zaragoza, Spain